CLINICAL TRIAL: NCT03186131
Title: Examination of Bone Metabolism and Bone Mineral Density in Primary and Secondary Osteoporosis Treated by Oral Ibandronate
Brief Title: Efficacy of Oral Ibandronate in Osteoporosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Associate professor at Shinshu University, Shinshu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Oral IBN2017
Record Dates: First submitted 2017-06-05; First posted 2017-06-14 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Ibandronic Acid; Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Ibandronate alone (Active Comparator): Monthly Oral Intake of Ibandronate
  Interventions: Drug: Ibandronate
- Oral Ibandronate and Vitamin D (Active Comparator): Monthly oral intake of Ibandronate and daily oral intake of Vitamin D
  Interventions: Drug: Oral Ibandronate and Vitamin D

INTERVENTIONS:
Drug: Ibandronate — To examine the efficacy of oral Ibandronate in osteoporosis
  Arms: Oral Ibandronate alone
Drug: Oral Ibandronate and Vitamin D — To examine the efficacy of oral Ibandronate and Vitamin D in osteoporosis
  Arms: Oral Ibandronate and Vitamin D

SUMMARY:
There has been no comparative data between oral ibandronate and oral ibandronate plus active vitamin D

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic patients who want to take oral ibandronate

Exclusion Criteria:

* Patients who are allergic to oral ibandronate or vitamin D Patients who have not taken oral ibandronate for the last 2 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients are separately analyzed
Enrollment: 100 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2022-12-08 (Estimated); Study Completion 2025-06-08 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | Change from Baseline Values at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No